CLINICAL TRIAL: NCT03184519
Title: Comparison of hhCG With hCG+ß in the Early Prediction of Ongoing Pregnancy After In-vitro Fertilization and Embryo Transfer.
Brief Title: Comparison of hhCG With hCG+ß in the Early Prediction of Ongoing Pregnancy.
Acronym: hyperPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1701-VLC-011-EB
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Results first posted 2020-03-04 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Pregnancy Test
MeSH Terms: interventions — Pregnancy Tests

STUDY DESIGN:
Intervention Model Description: All the patients will undergo 3 blood samples for analyses to determine pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Patients will undergo 3 blood samples after IVF-ET (pregnancy test) to determine pregnancy.
  Interventions: Diagnostic Test: Pregnancy test

INTERVENTIONS:
Diagnostic Test: Pregnancy test — Instead of one blood sample, patients will have three blood analyses to predict pregnancy earlier after the embryo transfer.

SUMMARY:
Proof of concept study for the prediction of ongoing pregnancy in women undergoing In-Vitro Fertilization (IVF), using hyperglycosylated human chorionic gonadotropin (hhCG), early after In-Vitro Fertilization and fresh Embryo Transfer (IVF-ET).

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Patients undergoing their first or second IVF-ET cycle
* Age 18-45 years
* Use of Ovitrelle for final follicular maturation and luteinization
* Fresh or Frozen day-5 blastocysts transrer (Autologus or Egg donation)

Exclusion criteria:

* Gestational surrogacy (patient's eggs used for pregnancy in a surrogate mother)
* Canceled IVF cycles
* GnRH agonist triggering cycles in the case of fresh ET.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 156 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Bosch, MDPhD, Principal Investigator — IVIRMA VALENCIA
Locations (1):
- IVI Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 156
Completed | 129
Not Completed | 27
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 21

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 155
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 39 [27 to 45]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 155
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  hispanic/latino | 2
  not hispanic/latino | 153
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  CAUCASIAN | 155
  ARAB NORTH | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Early Detection of Pregnancy
Description: Detection of Pregnancy on earlier dates (before day-11 after Embrio transfer)
Time Frame: One month
Population: From the 155 patients, 13 were excluded from analysis for several issues.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 142
Participants | 142
Statistical Analysis 1: Comparison: All Patients; Test type: Superiority; p = 0.025, t-test, 1 sided; Area Under Curve = 0.79

ADVERSE EVENTS:
Time Frame: 10 MONTH
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/156
Serious Adverse Events (participants affected / at risk) | 0/156
Other Adverse Events (participants affected / at risk) | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT03184519/Prot_SAP_000.pdf